CLINICAL TRIAL: NCT04840342
Title: Role of LSD1 in Hypertension in Blacks
Brief Title: MR Antagonist and LSD1
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrea Haas, M.D., Principal Investigator, Instructor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021p000990
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Mineralocorticoid Excess
MeSH Terms: conditions — Hypertension; Hyperaldosteronism | interventions — Eplerenone; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eplerenone Arm (Experimental): We posit that individuals who carry the LSD1 risk allele have increased mineralocorticoid receptor activity, which results in hypertension. Thus, our mechanistic clinical study will assess whether hypertensive LSD1 risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine). To test this hypothesis, we will perform a randomized, double-blind, active controlled study in hypertensive carriers of the LSD1 risk allele using a novel two-limb, proof-of-principle study. Our primary outcome will be a liberal salt diet systolic blood pressure. Therefore, this mechanistic trial will provide support for using a genetic marker that identifies individuals who are uniquely responsive to mineralocorticoid receptor blockade--personalized, precision medicine.
  Interventions: Drug: Eplerenone
- Amlodipine Arm (Experimental): We posit that individuals who carry the LSD1 risk allele have increased mineralocorticoid receptor activity, which results in hypertension. Thus, our mechanistic clinical study will assess whether hypertensive LSD1 risk allele carriers will show significantly greater reductions in blood pressure with a specific aldosterone mediated treatment approach (mineralocorticoid receptor blockade) than with a non-specific approach (amlodipine). To test this hypothesis, we will perform a randomized, double-blind, active controlled study in hypertensive carriers of the LSD1 risk allele using a novel two-limb, proof-of-principle study. Our primary outcome will be a liberal salt diet systolic blood pressure. Therefore, this mechanistic trial will provide support for using a genetic marker that identifies individuals who are uniquely responsive to mineralocorticoid receptor blockade--personalized, precision medicine.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Eplerenone — Dose escalations of eplerenone 50, 100, or 200mg
  Arms: Eplerenone Arm
Drug: Amlodipine — Dose escalations of amlodipine 2.5, 5, or 10mg
  Arms: Amlodipine Arm

SUMMARY:
Lysine specific demethylase-1 (LSD1) is an epigenetic regulator of gene transcription involved in the pathophysiology of elevated blood pressure and likely renal damage in Blacks. This project investigates whether a genetically driven anti-hypertensive approach proves superior in controlling blood pressure and mitigating renal injury in Blacks who carry the risk allele for LSD1 (rs587168). The findings of these investigations may lead to a new approach in treating a subset (~30%) of the essential hypertension population (Black LSD1 risk allele hypertensives).

DETAILED DESCRIPTION:
This proof-of-principle physiologic study in hypertensive Black LSD1 risk allele carriers testing the hypothesis that reductions in blood pressure will be greater with a genetically-driven anti-hypertensive approach (mineralocorticoid receptor antagonist, eplerenone) compared to a non-specific approach (amlodipine). 56 participants will be enrolled in a 12-week randomized, double-blind, active controlled, outpatient study to assess whether eplerenone (LSD1 specific treatment) proves superior in 24-hr ambulatory systolic blood pressure reduction than amlodipine (non-specific treatment). Participants will be randomized to either eplerenone 50mg or amlodipine 2.5mg with escalations in dose of study drug every 4 weeks if the participant's blood pressure is > 140/90.

ELIGIBILITY:
Inclusion Criteria:

* untreated as well as currently treated hypertensives
* rs587168 allele carriers
* not on more than two anti-hypertensives
* normal renal, metabolic, electrolyte, and CBC laboratory tests
* self-identified Black race
* age >17 yrs.

Exclusion Criteria:

* known cardiac disease other than HTN
* renal, circulatory or neurologic diseases
* diabetes
* smoking
* secondary HTN as indicated by history, physical examination or screening blood and urine tests
* smoking
* any drug therapy, except for anti-hypertensives and stable thyroid medication replacement

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
24-hour systolic ambulatory blood pressure | Change in systolic blood pressure between baseline and 4 weeks on study drug
  Subjects will be counseled regarding liberal salt dietary intake to ensure similar intakes in all subjects [Na+ (200 mEq), potassium (K+, 100 mEq) and calcium (800 mg)]. After completion of this diet for 6 days, the subject will collect a 24-hour ambulatory blood pressure. Procedure will be performed before randomization and after 4 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Haas, MD, Principal Investigator — Brigham and Women's
Locations (1):
- Brigham and Women's, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No